CLINICAL TRIAL: NCT04843800
Title: Imaging Pain! Ultrasound-based Palpation and Visualization for Diagnosing Chronic Low Back Pain
Brief Title: Ultrasound of the Thoracolumbar Fascia for Diagnosing Chronic Low Back Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The grant money has been used up.
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CE 21.003; 2021-AUDC-284121 (Other Grant/Funding Number: Fonds de recherche du Québec)
Record Dates: First submitted 2021-04-07; First posted 2021-04-14 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Low Back Pain
Keywords: Ultrasound imaging; Elastography; Lumbar fascia; Acupuncture therapy; Manipulation, Chiropractic; Massage therapy
MeSH Terms: conditions — Low Back Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: The patients will be randomized in three groups (allocation 1:1). Group 1 will receive a standardized acupuncture treatment and Group 2 will receive a standardized chiropractic treatment. Both groups will receive one treatment session per week for 3 consecutive weeks. Following the third treatment, at week 4, the US exam will be repeated and the questionnaires will be administered again.
  Group 3 will be placed on a waiting list for 3 weeks and will be reexamined by US and respond to the questionnaires at week 4. Then the group 3 patients will undergo a standardized therapeutic massage treatment consisting of one treatment session per week for 3 consecutive weeks. Following the third treatment, at week 7, the US exam will be repeated and the questionnaires will be administered again.
Who Masked: Outcomes Assessor
Masking Description: Ultrasound data analysis will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture (Experimental): The acupuncture treatments will consist of one 45-minute session weekly, for 3 consecutive weeks. The acupuncture treatment protocol will be semi standardized according to usual practice. All patients will be treated with a selection of local and distant points, comprising 10 minutes of insertion time, 30 minutes of needle retention and manipulation to achieve de qi (an irradiating feeling) if possible.
  Interventions: Procedure: Manual therapy
- Chiropractic (Experimental): The chiropractic treatments will consist of one 20-minute session weekly, for 3 consecutive weeks. The Diversified technique is one of the most commonly practiced techniques by chiropractors. In the treatment of low back pain, this technique involves the application of a quick (high-velocity), short (low-amplitude) thrust (adjustment) to the lumbo-pelvic area.
  Interventions: Procedure: Manual therapy
- Waiting list and Therapeutic Massage (Experimental): The therapeutic massage treatments will consist of one 45-minute session weekly, for 3 consecutive weeks. A technique called Fascial Release will be used. Tension related to back pain is believed to be present not only in the back but also in various parts of the body such as the legs, through the connection of fascia, the membrane that surrounds the muscles. The purpose of this treatment is to reduce the tension connected to the lower back.
  Interventions: Procedure: Manual therapy

INTERVENTIONS:
Procedure: Manual therapy — Acupuncture, Chiropractic are recognized complementary medicines and Therapeutic Massage is an alternative healing practice.

SUMMARY:
It is estimated that 23% of Quebecers suffer from chronic low back pain, and that 12% are disabled by this condition. Despite medical advances, the origin of so-called 'nonspecific low back pain' remains enigmatic. Conventional imaging methods by computed tomography and magnetic resonance may provide information on vertebral structures. However, very often, they do not diagnose lesions that genuinely correlate with the patient's symptoms. The lack of accurate diagnosis limits the therapeutic management in these patients.

Therefore, patients are increasingly turning to alternative and complementary medicine therapies (e.g., acupuncture, chiropractic , osteopathy, shiatsu) to relieve their pain. These therapies target painful areas of abnormal hardening in muscles of the lower back and aim to release the tension in these tissues to control pain. However, these painful areas and their resolution after manual therapy have yet to be demonstrated by means other than manual palpation. We will conduct a randomized controlled trial in chronic low back pain patients to examine the effects of acupuncture, chiropractic therapy and therapeutic massage on lower back muscular and connective tissues' physical properties using innovative ultrasound techniques.

DETAILED DESCRIPTION:
This will be a phase II, prospective, randomized controlled study, which will have received IRB approval and will be registered at Clinicaltrials.gov before it begins. Participants with chronic non specific low back pain (NSLBP) will be recruited from one site. On the day of the registration visit, the participants will meet with the research assistant to review and sign the consent form, give clinical and demographic data and respond to validated outcome questionnaires.

The participants will then undergo a research dynamic ultrasound (US) of the lower back. One musculoskeletal radiologist will perform the US exams consisting of a series of 5 dynamic scans of both the right and left paraspinal muscles, obtained during passive flexion of the lower body. Following the US exam, the participants will be randomized in three groups (allocation 1:1). One group will receive a standardized acupuncture treatment and another group will receive a standardized chiropractic treatment. One treatment session per week for 3 consecutive weeks will be provided. Following the 3 treatment sessions, at week 4, the US exam will be repeated and the questionnaires will be administered.

The third group will be placed on a waiting list for 3 weeks and will be reexamined by US and respond to the questionnaires at week 4. Then, the participants will undergo a standardized therapeutic massage treatment with one treatment session per week for 3 consecutive weeks. Following the 3 treatment sessions, at week 7, the US exam will be repeated and the questionnaires will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Ongoing low back and/or referred pain (non-specific pattern) above or just below the gluteal fold of at least 3/10 on a numerical pain rating scale (NRS), for at least 3 months;
* Pain has resulted in a problem on at least 50% of the days in the past 6 months;
* Only use of oral non-steroidal anti-inflammatory drugs for pain treatment in the 4 weeks before treatment;
* Willingness to commit to treatment sessions (acupuncture, chiropractic therapy or therapeutic massage) and to follow-up visits.

Exclusion Criteria:

* Back pain attributable to a specific, recognizable, known pathology:

  1. protrusion or prolapse of 1 or more intervertebral discs with concurrent neurological symptoms;
  2. radicular pain (sciatica);
  3. infectious spondylopathy;
  4. low back pain caused by inflammatory, malignant, or autoimmune disease;
  5. congenital deformation of the spine (except for slight lordosis or scoliosis);
  6. compression fracture caused by osteoporosis;
  7. spinal stenosis;
  8. spondylolysis or spondylolisthesis;
  9. Pregnancy;
* History of spinal surgery;
* History of pelvis or hip fractures;
* Acupuncture, spinal manipulation or therapeutic massage for back pain within the past year;
* Severe clotting disorders or anticoagulant therapy;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
% shear strain change. | Change from baseline % shear strain at week 4 (Groups 1, 2 and 3). Change from week-4 % shear strain at week 7 (Group 3).
  Percent shear strain between the thoracolumbar fascia and the epimysium of the erector spinae muscle.

SECONDARY OUTCOMES:
Quantitative ultrasound marker 'μ' change. | Change from baseline marker 'μ' at week 4 (Groups 1, 2 and 3). Change from week-4 marker 'μ' at week 7 (Group 3)
  Statistical analysis of the echo envelope: the mean intensity μ. This marker is unitless.
Quantitative ultrasound marker 'α' change. | Change from baseline marker 'α' at week 4 (Groups 1, 2 and 3). Change from week-4 marker 'α' at week 7 (Group 3)
  Statistical analysis of the echo envelope: the scatterer clustering parameter α. This marker is unitless.
Quantitative ultrasound marker 'κ' change. | Change from baseline marker 'κ' at week 4 (Groups 1, 2 and 3). Change from week-4 marker 'κ' at week 7 (Group 3)
  Statistical analysis of the echo envelope: the structure parameter κ. This marker is unitless.
Brief Pain Inventory short form 'pain severity' change. | Change from baseline BPI-sf pain severity at week 4 (Groups 1, 2 and 3). Change from week-4 BPI-sf pain severity at week 7 (Group 3)
  The Brief Pain Inventory short form (BPI-sf) is a self-administered questionnaire used to assess the severity of a patient's pain and the impact of this pain on the patient's daily functioning. The BPI-sf includes the four pain severity items (worst pain in last 24 hours, least pain in last 24 hours, pain on average, pain right now) and the seven interference items (general activity; mood; walking ability; normal work including housework; relations with other people; sleep; enjoyment of life). Each item is scored on an 11-point numerical rating scale (NRS) where 0 indicates no pain and 10 indicates worst pain imaginable. There is no scoring algorithm. The arithmetic mean of the four severity items will be used as measures of pain severity; the arithmetic mean of the seven interference items will be used as a measure of pain interference. The minimum and maximum values are 0 and 10 respectively. A higher score represents a worse outcome.
Brief Pain Inventory short form 'pain interference' change. | Change from baseline BPI-sf pain interference at week 4 (Groups 1, 2 and 3). Change from week-4 BPI-sf pain interference at week 7 (Group 3)
  The Brief Pain Inventory short form (BPI-sf) is a self-administered questionnaire used to assess the severity of a patient's pain and the impact of this pain on the patient's daily functioning. The BPI-sf includes the four pain severity items (worst pain in last 24 hours, least pain in last 24 hours, pain on average, pain right now) and the seven interference items (general activity; mood; walking ability; normal work including housework; relations with other people; sleep; enjoyment of life). Each item is scored on an 11-point numerical rating scale (NRS) where 0 indicates no pain and 10 indicates worst pain imaginable. There is no scoring algorithm. The arithmetic mean of the four severity items will be used as measures of pain severity; the arithmetic mean of the seven interference items will be used as a measure of pain interference. The minimum and maximum values are 0 and 10 respectively. A higher score represents a worse outcome.
Oswestry Disability Index (ODI) change. | Change from baseline ODI at week 4 (Groups 1, 2 and 3). Change from week-4 ODI at week 7 (Group 3)
  Self-administered questionnaire. This test is widely used as a low back functional outcome tool. The minimum and maximum values are 0% and 100% respectively. A higher score means a worse outcome.
PROMIS (Patient-Reported Outcomes Measurement Information System) Global Health Scale change. | Change from baseline PROMIS Global Health at week 4 (Groups 1, 2 and 3). Change from week-4 PROMIS Global Health at week 7 (Group 3)
  Self-administered questionnaire. The PROMIS uses T scores. A score of 50 represents the mean of the concepts being measured, in the reference population. The standard deviation is 10. The range is from 0 to 100. Higher scores equals more of the concept being measured, therefore a better global health.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie J Bureau, MD MSc, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No